CLINICAL TRIAL: NCT07075094
Title: Determination of the Effectiveness of Two Different Noninvasive Stimulation Methods in Urine Collection in Infants: A Randomized Controlled Trial
Brief Title: Determination of the Effectiveness of Two Different Noninvasive Stimulation Methods in Urine Collection in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-01/77
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Infant; Urine; Nursing Interventions
Keywords: Infant; Urine collection; Noninvasive stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to experimental and control groups using block randomization method. Age and sex variables will be used for block randomization. In order to reach the sample size calculated in the study, strata will be repeated two times (2X2X6) and 24 infant will be included in each group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Using the block randomization technique, participants will be divided into 3 groups. A web-based randomization list creation tool will be used to create the blocked randomization list. Control and intervention groups will be coded as A, B and C using the sealed envelope method. Randomization information will be kept from the researcher involved in data collection until data collection begins. The researcher will learn which group each child is in just before the application (researcher blinding).Research data will be entered into the computer database by coding the group name as A, B and C, and statistical analysis will be performed using this coding (statistician blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Urine samples from infants in the control group will be collected according to the clinic's routine practice. Unlike routine practice, these infants will be positioned to ensure similarity to the experimental groups. Urine samples will be collected in an upright position, held under the arms. No noninvasive stimulation will be used.
- Bladder stimulation (Experimental): These babies will be held in an upright position by holding them under their arms during the urine sample collection process. A bladder stimulation technique will be used during the procedure.
  Interventions: Procedure: Bladder stimulation
- Subrapubic cutaneous stimulation (Experimental): These babies will be held in an upright position by holding them under their arms during the urine sample collection process. A subrapubic cutaneous stimulation technique will be used during the procedure.
  Interventions: Procedure: Subrapubic cutaneous stimulation

INTERVENTIONS:
Procedure: Bladder stimulation — This stimulation consists of two stages. In the first maneuver, the bladder is stimulated by gentle tapping of the suprapubic area for 30 seconds. In the second maneuver, the paravertebral area is massaged in a circular motion for 30 seconds. The two stimulation maneuvers are repeated sequentially for 5 minutes.
  Arms: Bladder stimulation
Procedure: Subrapubic cutaneous stimulation — Circular rubbing movements will be made on the baby's suprapubic area with gauze soaked in cold salt water until micturition begins.
  Arms: Subrapubic cutaneous stimulation

SUMMARY:
This study will be conducted to determine the effects of bladder stimulation and subrapubic cutaneous stimulation techniques applied during urine sampling in infants on the success of urine sampling, pain and procedure time.

DETAILED DESCRIPTION:
Urinary tract infections are common in children. Urine samples and urinalysis are needed to confirm the diagnosis of urinary tract infection. Various invasive and noninvasive techniques are used for urine sample collection in children. These techniques include suprapubic aspiration, urinary catheterization, a sterile urine bag, and clean catch techniques. The clean catch technique is a commonly used noninvasive technique for urine sample collection in children. Parents have described clean catch urine collection in children who are not toilet-trained as time-consuming and complex. Alternative techniques that stimulate voiding in children who are not toilet-trained, allowing for quicker collection of urine samples using clean catch techniques, are beneficial. The noninvasive stimulation methods whose effectiveness in infant urine collection will be evaluated in this study are bladder stimulation and suprapubic cutaneous stimulation.

ELIGIBILITY:
Inclusion Criteria:

* A urine sample must be collected due to suspicion of a urinary tract infection,
* The infant must be being fed orally,
* The skin in the area where the maneuver will be performed must be intact,
* The infant must be conscious and have stable vital signs.
* The infant must be from families that can speak and understand Turkish and are willing to participate in the study

Exclusion Criteria:

* Presence of respiratory distress and signs of dehydration,
* Presence of a diagnosed chronic health problem,
* Presence of a neurological or anatomical abnormality that may affect bladder function,
* Presence of any diagnostic suspicion (distension, intussusception, appendicitis, etc.) that would preclude the application of the stimulation maneuver,
* Presence of cold stress.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Procedural pain score- FLACC Pain Scale | At the beginning of the procedure, at the end of the procedure
  The Face, Legs, Activity, Cry, and Consolability (FLACC) scale consists of five categories (face, legs, activity, crying, and consolability), and each category is scored between 0 and 2 depending on the pain or distress behaviors observed. The total score ranges from 0 to 10, with 0 indicating no pain or distress and 10 indicating extreme pain or distress. The FLACC scale was developed to assess pain in children aged 2 months to 7 years and is one of the widely recommended scales for assessing pain and distress among pediatric patients.
Urine sample collection success | During the procedure (Average 5 minutes)
  Infants who can have a urine sample collected during the procedure will be recorded as having a successful procedure.

SECONDARY OUTCOMES:
Procedure time | Through the procedure completion, an average of 5 minutes.
  Procedure time is the time between the start of the stimulation method and the start of micturition.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Ozdemir, Professor, Study Director — İstanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: January through March of 2027
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Marchal S, Janicot J, Salicis J, Demonchy D, Herisse AL, Olla M, Rancurel A, Haas H, Berard E, Breaud J, Bernardor J, Ribet C, Freyssinet E, Donzeau D, Desmontils J, Schori-Fortier C, Fontas E, Tran A. Quick-Wee versus bladder stimulation to collect midstream urine from precontinent infants under 1 year of age: a study protocol for a randomised controlled trial (ES.Stimquick.U). BMJ Open. 2021 Sep 16;11(9):e046324. doi: 10.1136/bmjopen-2020-046324. PMID 34531206
- [Background] Korkmaz N, Narter FK, Mutlu B, Sahin K, Ozgoru H. Effects of the bladder stimulation technique on urine sample collection in newborns: A randomized controlled study. Int J Nurs Pract. 2024 Oct;30(5):e13255. doi: 10.1111/ijn.13255. Epub 2024 Apr 15. PMID 38622105